CLINICAL TRIAL: NCT03399526
Title: A 28-day, Double-blind, Randomized, Reference-controlled Open Psoriasis Plaque Test for Within Subject Comparison of Efficacy and Safety of Mapracorat 0.1% Ointment and 4 Reference Products in Symptomatic Volunteers With Stable Plaque-type Psoriasis
Brief Title: 1404003_OpenPsori.PlaqueTest to Eval.Eff.of Diff.Comp. to Mapracorat
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16599; 2012-004171-39 (EudraCT Number)
Record Dates: First submitted 2018-01-09; First posted 2018-01-16 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2017-12

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — R-1,1,1-trifluoro-4-(5-fluoro-2,3-dihydrobenzofuran-7-yl)-4-methyl-2-(((2-methyl-5-quinolyl)amino)methyl)pentan-2-ol; prednicarbate; Ointments; Clobetasol; calcipotriene; betamethasone-17,21-dipropionate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Mapracorat (Experimental): 10 µL of mapracorat was applied on 6 days a week for up to 4 weeks onto the corresponding test fields (3 cm2) of the affected skin plaques (15 cm2 were treated in total [diameter 2 cm, distance to next test field at least 2 cm]). 200 µL of mapracorat was applied on 6 days a week for up to 4 weeks onto the defined test fields (12.5 cm2 were treated in total [diameter 1.8 cm, distance to next test field at least 1.5 cm]) occluded with Finn chambers of the non-lesional skin areas of 2.5 cm2
  Interventions: Drug: Mapracorat (ZK 245186, BAY 86-5319)
- Prednicarbate (Active Comparator): 10 µL of prednicarbate was applied on 6 days a week for up to 4 weeks onto the corresponding test fields (3 cm2) of the affected skin plaques (15 cm2 were treated in total [diameter 2 cm, distance to next test field at least 2 cm]). 200 µL of prednicarbate was applied on 6 days a week for up to 4 weeks onto the defined test fields (12.5 cm2 were treated in total [diameter 1.8 cm, distance to next test field at least 1.5 cm]) occluded with Finn chambers of the non-lesional skin areas of 2.5 cm2
  Interventions: Drug: Prednicarbate 0.25% ointment
- Clobetasol (Active Comparator): 10 µL of clobetasol was applied on 6 days a week for up to 4 weeks onto the corresponding test fields (3 cm2) of the affected skin plaques (15 cm2 were treated in total [diameter 2 cm, distance to next test field at least 2 cm]). 200 µL of clobetasol was applied on 6 days a week for up to 4 weeks onto the defined test fields (12.5 cm2 were treated in total [diameter 1.8 cm, distance to next test field at least 1.5 cm]) occluded with Finn chambers of the non-lesional skin areas of 2.5 cm2
  Interventions: Drug: Clobetasol 0.05% ointment
- Calcipotriene (Active Comparator): 10 µL of calcipotriene was applied on 6 days a week for up to 4 weeks onto the corresponding test fields (3 cm2) of the affected skin plaques (15 cm2 were treated in total [diameter 2 cm, distance to next test field at least 2 cm]). 200 µL of calcipotriene was applied on 6 days a week for up to 4 weeks onto the defined test fields (12.5 cm2 were treated in total [diameter 1.8 cm, distance to next test field at least 1.5 cm]) occluded with Finn chambers of the non-lesional skin areas of 2.5 cm2
  Interventions: Drug: Calcipotriene 0.005% ointment
- Calcipotriene/Betamethasone dipropionate (Active Comparator): 10 µL of calcipotriene/betamethasone dipropionate was applied on 6 days a week for up to 4 weeks onto the corresponding test fields (3 cm2) of the affected skin plaques (15 cm2 were treated in total [diameter 2 cm, distance to next test field at least 2 cm]). 200 µL of calcipotriene/betamethasone dipropionate was applied on 6 days a week for up to 4 weeks onto the defined test fields (12.5 cm2 were treated in total [diameter 1.8 cm, distance to next test field at least 1.5 cm]) occluded with Finn chambers of the non-lesional skin areas of 2.5 cm2
  Interventions: Drug: Calcipotriene 0.005%/Betamethasone dipropionate 0.05% ointment

INTERVENTIONS:
Drug: Mapracorat (ZK 245186, BAY 86-5319) — 0.1% (1 mg/g) of the active ingredient mapracorat plus excipients as ointment
  Arms: Mapracorat
Drug: Prednicarbate 0.25% ointment — 0.25% (2.5 mg/g) of the active ingredient prednicarbate as ointment
  Arms: Prednicarbate
Drug: Clobetasol 0.05% ointment — 0.05% (0.5 mg/g) of the active ingredient clobetasol as ointment
  Arms: Clobetasol
Drug: Calcipotriene 0.005% ointment — 0.005% (0.05 mg/g) of the active ingredient calcipotriene as ointment
  Arms: Calcipotriene
Drug: Calcipotriene 0.005%/Betamethasone dipropionate 0.05% ointment — 0.005% (0.05 mg/g) of the active ingredient calcipotriene/0.05% (0.5 mg/g) of the active ingredient betamethasone dipropionate as ointment
  Arms: Calcipotriene/Betamethasone dipropionate

SUMMARY:
Evaluation of efficacy and safety of Mapracorat 0.1% ointment and 4 comparator ointments in male and female subjects 18 to 65 years with stable plaque-type psoriasis treated once daily 6 days a week for a maximum of 4 weeks.

Primary objective was to compare the efficacy of all test compounds by measurement of psoriatic infiltrate thickness (PIT) with 20 MHz B mode ultrasound.

Secondary objectives were to assess safety of all test compounds by measurement of the atrophogenic potential on non-lesional skin with 20 MHz B mode ultrasound, to assess the efficacy of all test compounds by measurement of intensity of erythema measured by chromametry, to assess the efficacy of all test compounds by visual assessment of the skin in the test fields using a 5-point score, to assess the safety of all test compounds by visual assessments of formation of teleangiectasia using a 5-point score, to assess the safety of all test compounds by visual assessment of atrophy using a 5-point score, to assess the safety of all test compounds by visual assessment of local tolerability using a 5-point score, to visualize the therapeutic index given by PIT versus non lesional skin thickness.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18 to 65 years of age with stable plaque-type psoriasis, plaques of adequate size to allow for evaluation of 5 test fields, on comparable body area; thickness of the echo-lucent band under the entry echo as assessed by ultrasound of at least 200 μm

Exclusion Criteria:

* Positive testing in urine drug screening
* Pregnancy or lactation
* A history of relevant diseases, especially-incompletely cured pre-existing diseases for which it could have been assumed that the absorption, distribution, excretion and effect of the study drugs would not be normal
* Volunteers with severe kidney or liver disease
* Volunteers with concurrent/acute viral infections in the test field areas (e.g. herpes simplex, varicella) or other specific skin alterations (skin tuberculosis, syphilitic skin lesions)
* Severe disease within the last 4 weeks prior to the first study drug administration
* Volunteers with known hypersensitivity reaction when applying adhesive bandages
* Volunteers who were treated with any systemic therapy for psoriasis (e.g. methotrexate, cyclosporin A, etretinate, acitretin, PUVA, fumaric acid) three months prior to screening
* Volunteers who were treated with any systemic corticosteroids (oral, intramuscular, high-dose inhaled, rectal) 4 weeks prior to screening
* Volunteers who were treated with any local therapy for psoriasis (e.g. corticosteroids, calcitriol analogues, dithranol, phototherapy) 2 weeks prior to screening
* Target plaques localized on head and neck, elbows and knees, palms and soles, nails and folds or other mechanically strained sites
* Volunteers with guttate or pustular psoriasis
* Volunteers with spontaneously improving or rapidly deteriorating plaque-type psoriasis
* Volunteers with erythrodermic type of psoriasis
* Volunteers with severe recalcitrant psoriasis requiring additional therapy
* Presence of hepatitis B virus surface antigen, hepatitis C virus antibodies or human immune deficiency virus antibodies
* Clinico-chemical parameters of clinically significant deviation
* Volunteers with a known allergy to any of the excipients of the trial medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-02-11 (Actual); Primary Completion 2013-05-31 (Actual); Study Completion 2013-05-31 (Actual)

PRIMARY OUTCOMES:
Baseline-corrected area under the curve of the psoriatic infiltrate thickness (PIT) measured by 20 MHz B mode ultrasound | Prior to drug application from Day 1 and up to Day 29
  Assessment was done on the test fields on psoriatic plaques

SECONDARY OUTCOMES:
Skin thickness measurement of occluded test field on non-lesional skin (mean of triplicate measurement) | Prior to drug application from Day 1 up to Day 60
  Assessment was made on occluded test fields on non-lesional skin areas on the forearm
Clinical assessment of atrophy using a 5-point score | Prior to drug application from Day 1 and up to Day 29
  Assessment was made on occluded test fields on non-lesional skin areas on the forearm
Clinical assessment of telangiectasia using a 5-point score | Prior to drug application from Day 1 and up to Day 29
  Assessment was made on occluded test fields on non-lesional skin areas on the forearm
Clinical assessment of local tolerability using a 5-point score | Prior to drug application from Day 1 and up to Day 29
  Assessment was made on occluded test fields on non-lesional skin areas on the forearm
PIT measured by 20 MHz B mode ultrasound | Prior to drug application from Day 1 and up to Day 29
  Assessment was done on the test fields on psoriatic plaques
Measurement of erythema using chromametry (mean of triplicate measurement) | Prior to drug application from Day 1 and up to Day 29
  Assessment was done on the test fields on psoriatic plaques
Clinical efficacy assessment of the skin in the test fields using a 5-point score | Prior to drug application from Day 1 and up to Day 29
  Assessment was done on the test fields on psoriatic plaques
Number of participants with adverse events | Approximately 64-84 days

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Hamburg, Germany

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/